CLINICAL TRIAL: NCT02583789
Title: A Double-blinded, Placebo-controlled, Crossover Study to Assess Efficacy of Oral Treprostinil Titrated to Highest Tolerable Dose in 20 Patients With Symptomatic Primary or Secondary Raynaud's Phenomenon Resistant to Vasodilatory Therapy
Brief Title: Assess Efficacy of of Oral Treprostinil in Patients With Symptomatic Primary or Secondary Raynaud's Phenomenon
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Principal Investigator, Aaron Waxman MD PhD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015P001879
Record Dates: First submitted 2015-10-08; First posted 2015-10-22 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Raynaud's Phenomenon
MeSH Terms: conditions — Raynaud Disease | interventions — treprostinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral treprostinil (Active Comparator): Dosing of oral treprostinil will be initiated at 0.125 mg three times daily. Dose escalations of oral treprostinil can occur every 72 hours (three consecutive doses) in 0.125 mg increments. Subjects will be titrated as tolerated to a goal dose of 2mg TID over a 6-week period.
  Interventions: Drug: oral treprostinil; Drug: Placebo
- Placebo (Placebo Comparator): Placebo mimics oral treprostinil and will be taken three times a day
  Interventions: Drug: oral treprostinil; Drug: Placebo

INTERVENTIONS:
Drug: oral treprostinil — Change in the Raynaud's Condition Score from baseline (2-week run in), comparing treprostinil treatment phase vs. placebo phase
  Other Names: Orenitram
Drug: Placebo — Placebo is a sugar pill manufactured to resemble UT-15C. Change in the Raynaud's Condition Score from baseline (2-week run in), comparing treprostinil treatment phase vs. placebo phase
  Other Names: Sugar pill

SUMMARY:
This study represents the first trial to assess the efficacy of oral treprostinil therapy in patients with symptomatic primary or secondary Raynaud's Phenomenon (RP) resistant to vasodilatory therapy.

The study will be randomized 1:1 UT-15C to placebo. The design is a crossover study and all subjects will be randomized to receive oral treprostinil sustained release tablets or matching placebo for 12 weeks and then crossover for 12 weeks. All subjects will be exposed for 12 weeks of treatment with oral UT-15C during the study.

DETAILED DESCRIPTION:
A single center double-blinded, placebo-controlled, crossover study to assess efficacy of oral treprostinil titrated to a tolerable goal dose of 2.0 mg three times per day (TID) in 20 patients with symptomatic primary or secondary Raynaud's Phenomenon resistant to vasodilatory therapy. Based on a pre-screening survey of the clinic population we anticipate at least 30 patients per year will be eligible for enrollment. At the clinicians discretion the dose can be increased as tolerated.

Eligible subjects at the time of signing an informed consent will have a diagnosis of primary or secondary Raynaud's Phenomenon. Subjects will be recruited from the Raynaud's Clinic, which is a multidisciplinary clinic held at the Watkins Clinic at the Shapiro Cardiovascular Center. Subjects will be assessed during a Screening and treatment initiation visit to determine eligibility for the study.

This study represents the first trial to assess the efficacy of oral treprostinil therapy in patients with symptomatic primary or secondary Raynaud's phenomenon resistant to vasodilatory therapy.

Oral treprostinil (UT-15C), a synthetic prostacyclin analog that inhibits platelet aggregation, induces vasodilation, and suppresses smooth muscle proliferation. In a recent open label study of escalating doses of oral treprostinil in patients with systemic sclerosis and digital ischemia, oral treprostinil was effectively absorbed in patients with scleroderma and was temporally associated with improved cutaneous perfusion and temperature. Thus, oral treprostinil may provide a new therapeutic option for patients with refractory secondary Raynaud's Phenomenon.

A recent systematic review demonstrated that oral calcium channel blockers, the most commonly prescribed drugs for primary RP, are only minimally effective in reducing the frequency of attacks and severity. Although Sildenafil has been shown to increase digital skin blood flow during all phases of local cooling in primary RP, its role in primary RP is not yet confirmed in randomized, controlled trials. To our knowledge, very few studies have assessed the use of oral prostacyclin therapy for disabling primary RP, although one multicenter, double-blind, randomized trial of an oral analog of prostacyclin, known as beraprost, reduced the number of RP attacks but proved no more beneficial than placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18-65 years
* Active Raynaud's Phenomenon defined as patients with refractory RP having four or more RP attacks per week in the 2 weeks before inclusion in the study despite treatment with vasodilators for at least 3 months
* Patients with primary Raynaud's Phenomenon
* Patients with Raynaud's secondary to connective tissue diseases (including scleroderma (SSc), limited scleroderma (CREST), mixed connective tissue disease (MCTD), primary Sjogren's syndrome (SS), systemic lupus erythematosus (SLE), with diagnosis of the underlying rheumatic disease based on standard criteria
* Patients on stable dose phosphodiesterase inhibitors (sildenafil, tadalafil or vardenafil), endothelin antagonists, alpha adrenergic antagonists, or calcium channel blockers defined as 3-months with no change in dose will be allowed to participate

Exclusion Criteria:

* Uncontrolled hypertension, diabetes mellitus, history of orthostatic hypotension, acute coronary or cerebrovascular event within 3 months, evidence of malignancy, history of sympathectomy
* Smoking within 3 months or smoking cessation using nicotine products
* Subjects currently taking or other prostacyclins.
* Pregnant or breast feeding or considering pregnancy in next 4 months
* Participation in trial with an investigational drug within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Raynaud's Condition Score | from baseline (2-week run in) to 6 weeks of treatment
  Change in the Raynaud's Condition Score from baseline (2-week run in), comparing treprostinil treatment phase vs. placebo phase

SECONDARY OUTCOMES:
Change in number of Raynaud's Phenomenon attacks | from baseline (2-week run in) to 6 weeks of treatment
  Change in the number of Raynaud's Phenomenon attacks per week during the sixth week of treatment phase compared to the number of Raynaud's Phenomenon attacks per week at baseline.
Change in duration of Raynaud's Phenomenon attacks | from baseline (2-week run in) to 6 weeks of treatment
  Change in the total duration of Raynaud's Phenomenon attacks per week during the sixth week of treatment compared to the total duration of Raynaud's Phenomenon attacks per week at baseline.
Reduction of ulcer burden among secondary Raynaud's Phenomenon patients | from baseline (2-week run in) to 6 weeks of treatment
  Decrease ulcer burden in secondary Raynaud's Phenomenon patients by reducing the time to heal active ulcers and/or reducing the number of new ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Waxman, MD/PhD, Principal Investigator — Brigham and Womens Hospital; Paul Dellaripa, MD, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ennis H, Hughes M, Anderson ME, Wilkinson J, Herrick AL. Calcium channel blockers for primary Raynaud's phenomenon. Cochrane Database Syst Rev. 2016 Feb 25;2(2):CD002069. doi: 10.1002/14651858.CD002069.pub5. PMID 26914257
- [Background] Roustit M, Hellmann M, Cracowski C, Blaise S, Cracowski JL. Sildenafil increases digital skin blood flow during all phases of local cooling in primary Raynaud's phenomenon. Clin Pharmacol Ther. 2012 May;91(5):813-9. doi: 10.1038/clpt.2011.302. Epub 2012 Mar 28. PMID 22453196
- [Background] Vayssairat M. Controlled multicenter double blind trial of an oral analog of prostacyclin in the treatment of primary Raynaud's phenomenon. French Microcirculation Society Multicentre Group for the Study of Vascular Acrosyndromes. J Rheumatol. 1996 Nov;23(11):1917-20. PMID 8923366